CLINICAL TRIAL: NCT04399707
Title: Transcutaneous Electrical Nerve Stimulation for Post-Cesarean Pain Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawaii Pacific Health (Other)
Responsible Party: Principal Investigator, Kelly Yamasato, MD, Physician, Assistant Professor, Hawaii Pacific Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-035
Record Dates: First submitted 2020-02-18; First posted 2020-05-22 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Transcutaneous Electric Nerve Stimulation; Analgesia; Cesarean Section
Keywords: TENS; Transcutaneous electric nerve stimulation; Cesarean analgesia
MeSH Terms: conditions — Agnosia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of three groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Active TENS Unit (Active Comparator)
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS) unit
- Placebo TENS Unit (Placebo Comparator)
  Interventions: Device: Placebo transcutaneous electrical nerve stimulation (TENS) unit
- No TENS Unit (No Intervention)

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) unit — Patients will be randomized to active TENS unit, placebo TENS unit, or no TENS unit
  Arms: Active TENS Unit
Device: Placebo transcutaneous electrical nerve stimulation (TENS) unit — Patients will be randomized to active TENS unit, placebo TENS unit, or no TENS unit
  Arms: Placebo TENS Unit

SUMMARY:
Purpose of study is to evaluate the efficacy of transcutaneous electrical nerve stimulation (TENS) for post-operative pain control after a cesarean delivery compared to placebo and no TENS.

ELIGIBILITY:
Inclusion Criteria:

- Women undergoing scheduled or non-urgent cesarean section

Exclusion Criteria:

* Non-English speaking
* Subjects with a history of chronic pain or chronic opioid use
* Pre-operative use of opioids for more than 1 week in the preceding 6 months
* Previous exposure to the TENS unit
* Women with an allergy or contraindication to narcotics/NSAIDs/acetaminophen
* Subjects who had a midline vertical skin incision during this operation
* Subjects who did not receive intrathecal opioids at the time of their cesarean delivery
* Adhesive allergies
* Subjects with a pacemaker (due to the unknown effects of the TENS on the electrical activity of the heart)
* Intraoperative general anesthesia
* Inability to consent to the study
* Postpartum tubal ligation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Post-operative narcotic consumption | First 60 hours post-operatively
  Total postoperative narcotic consumption (measured in morphine equivalents)

SECONDARY OUTCOMES:
Duration of hospitalization | From date of cesarean delivery until discharge from hospital, assessed up to 1 month
  Length of stay in hospital
Pain assessed by numeric analog scale (NAS) (0-10; 0: no pain at all, 10: worst imaginable pain) | On post-operative days 1, 2, 3, and day of discharge, assessed up to 1 month
  Pain scoring
Satisfaction with pain control assessed by NAS (0-10; 0: very dissatisfied, 10: very satisfied) | On post-operative days 1, 2, 3, and day of discharge, assessed up to 1 month
  Pain control satisfaction
Adverse reactions to TENS unit | From date of randomization until date of discharge, assessed up to 1 month
  Adverse reactions to TENS unit

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Yamasato, Principal Investigator — Physician
Locations (1):
- Nicole Kurata, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bateman BT, Franklin JM, Bykov K, Avorn J, Shrank WH, Brennan TA, Landon JE, Rathmell JP, Huybrechts KF, Fischer MA, Choudhry NK. Persistent opioid use following cesarean delivery: patterns and predictors among opioid-naive women. Am J Obstet Gynecol. 2016 Sep;215(3):353.e1-353.e18. doi: 10.1016/j.ajog.2016.03.016. Epub 2016 Mar 17. PMID 26996986
- [Background] Desantana JM, Sluka KA, Lauretti GR. High and low frequency TENS reduce postoperative pain intensity after laparoscopic tubal ligation: a randomized controlled trial. Clin J Pain. 2009 Jan;25(1):12-9. doi: 10.1097/AJP.0b013e31817d1070. PMID 19158541
- [Background] Bjordal JM, Johnson MI, Ljunggreen AE. Transcutaneous electrical nerve stimulation (TENS) can reduce postoperative analgesic consumption. A meta-analysis with assessment of optimal treatment parameters for postoperative pain. Eur J Pain. 2003;7(2):181-8. doi: 10.1016/S1090-3801(02)00098-8. PMID 12600800
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Dowswell T, Bedwell C, Lavender T, Neilson JP. Transcutaneous electrical nerve stimulation (TENS) for pain relief in labour. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007214. doi: 10.1002/14651858.CD007214.pub2. PMID 19370680
- [Derived] Kurata NB, Ghatnekar RJ, Mercer E, Chin JM, Kaneshiro B, Yamasato KS. Transcutaneous Electrical Nerve Stimulation for Post-Cesarean Birth Pain Control: A Randomized Controlled Trial. Obstet Gynecol. 2022 Aug 1;140(2):174-180. doi: 10.1097/AOG.0000000000004798. Epub 2022 Jul 6. PMID 35852266